CLINICAL TRIAL: NCT02001077
Title: Sleep and Pain Interventions in Fibromyalgia: Hyperalgesia and Central Sensitization
Brief Title: Sleep and Pain Interventions in Fibromyalgia
Acronym: SPIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 627-2007; R01AR055160 (NIH)
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Insomnia; Fibromyalgia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fibromyalgia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CBT-I (Active Comparator): Participants will complete 8 weekly therapy sessions focused on improving sleep. A multicomponent CBT-I (Cognitive Behavioral Therapy for Insomnia) protocol will involve: sleep hygiene, stimulus control, sleep restriction, relaxation, and cognitive restructuring.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
- CBT-P (Active Comparator): Participants will complete 8 weekly therapy sessions focused on improving pain. A multicomponent CBT-P (Cognitive Behavioral Therapy for Pain) protocol will involve: pain education, relaxation, activity pacing, and cognitive restructuring.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Pain (CBT-P)
- Waitlist Control (WLC) (No Intervention): Participants in the WLC group will not receive any treatment between the baseline and post-treatment assessments. After the final follow-up assessment, they will be offered the opportunity to receive therapy which combines aspects of both CBT-I and CBT-P.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
  Arms: CBT-I
Behavioral: Cognitive Behavioral Therapy for Pain (CBT-P)
  Arms: CBT-P

SUMMARY:
This is a single-center, randomized controlled trial study design. Enrolled participants had comorbid fibromyalgia and chronic insomnia. Participants were randomized to a behavioral intervention for pain, a behavioral intervention for insomnia, or a waitlist control. The study intervention period lasted eight weeks. The objective of the study is to examine the impact of two behavioral treatments on sleep and pain and to better understand what causes chronic pain and chronic sleep disturbance.

DETAILED DESCRIPTION:
Participants will be asked to review the informed consent and consent to the study prior to any study procedure.

There are six phases of this study: 1. a telephone interview, 2. an in-home single night sleep recording, 3. a two-week baseline period, 4. an 8-week treatment period, 5. a two-week follow-up period, and 6. another two week follow-up period 6-months after the treatment period.

During the telephone interview, participants will be asked question about their sleep and pain history. Participants with poor sleep will visit the University of Florida for a medical history and will be connected to a machine which will monitor their sleep. Participants will return home to sleep while still connected to the machine and will return the machine to the University of Florida the next day. A third visit will consist of completing questionnaires and measuring response to a range of temperatures. Participants will complete brief daily questionnaires and wear an actigraph (wristwatch-like device) that measures arm movements for two weeks.

Participants will then be randomized to one of three groups: a pain treatment group, an insomnia treatment group or a waitlist control group. Both treatments consist of weekly therapy sessions for 8 consecutive weeks. Participants assigned to waitlist control will be offered therapy at no cost at the end of the study. Throughout these 8 weeks, participants in all three groups will be asked to complete daily sleep diaries.

The study consists of two follow-up periods consisting of two weeks, during which participants will wear the actigraph and complete daily sleep diaries. Participants will travel to the University two times during each follow-up period. One follow-up period will occur immediately following treatment, and the other will occur approximately 6 months following treatment. During each follow-up period, the first visits will involve being connected to the machine that monitors their sleep. Participants will then return home with the machine to sleep in their own beds. The second of these visits will occur the following day and will involve the return of the machine, completion of questionnaires, and measurement of participants' responses to a range of temperatures applied to their arm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia
* Diagnosis of insomnia
* No sleep medications for at least 1 month, or stable on medications for at least 6 months
* Willing to be randomly assigned to a treatment
* Able to read and understand English

Exclusion Criteria:

* Sleep disorder other than insomnia
* Bipolar disorder
* Seizure disorder
* Severe untreated psychopathology
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2009-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in time spent awake during the night. | Change from baseline to the two study follow-ups (immediately and 3-months following treatment)
  The change in the time participants report spending awake during the night. Sleep will be measured with daily diaries and, means of the 14 days collected at baseline, immediately, and 6 months following treatment will be calculated.
Change in mood. | Change from baseline to the two follow-up periods (immediately and 3-months following treatment)
  The change in reported mood as assessed by questionnaires from baseline to immediately and 6 months following treatment.

SECONDARY OUTCOMES:
Change in self-report of pain experience. | Change from baseline to the two follow-up periods (immediately and 3-months following treatment)
  The change in participants' report of their pain experience from baseline to the two follow-up periods. Pain will be assessed by daily diaries, and means of the 14 days collected at baseline, immediately, and 6 months following treatment will be calculated.
Change in mood. | Change from baseline to the two follow-up periods (immediately and 3-months following treatment).
  The change in reported mood as assessed by questionnaires from baseline to immediately and 6 months following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christina S McCrae, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Anderson RJ, McCrae CS, Staud R, Berry RB, Robinson ME. Predictors of clinical pain in fibromyalgia: examining the role of sleep. J Pain. 2012 Apr;13(4):350-8. doi: 10.1016/j.jpain.2011.12.009. Epub 2012 Mar 3. PMID 22381437
- [Derived] McGovney KD, Curtis AF, McCrae CS. Actigraphic Physical Activity, Pain Intensity, and Polysomnographic Sleep in Fibromyalgia. Behav Sleep Med. 2023 Jul-Aug;21(4):383-396. doi: 10.1080/15402002.2022.2102009. Epub 2022 Jul 20. PMID 35856908
- [Derived] McCrae CS, Craggs JG, Curtis AF, Nair N, Kay D, Staud R, Berry RB, Robinson ME. Neural activation changes in response to pain following cognitive behavioral therapy for patients with comorbid fibromyalgia and insomnia: a pilot study. J Clin Sleep Med. 2022 Jan 1;18(1):203-215. doi: 10.5664/jcsm.9540. PMID 34310276
- [Derived] Miller MB, Curtis AF, Chan WS, Deroche CB, McCrae CS. Daily associations between sleep and opioid use among adults with comorbid symptoms of insomnia and fibromyalgia. J Clin Sleep Med. 2021 Apr 1;17(4):729-737. doi: 10.5664/jcsm.9002. PMID 33226334
- [Derived] McCrae CS, Curtis AF, Miller MB, Nair N, Rathinakumar H, Davenport M, Berry JR, McGovney K, Staud R, Berry R, Robinson M. Effect of cognitive behavioural therapy on sleep and opioid medication use in adults with fibromyalgia and insomnia. J Sleep Res. 2020 Dec;29(6):e13020. doi: 10.1111/jsr.13020. Epub 2020 Mar 3. PMID 32126156
- [Derived] Curtis AF, Miller MB, Rathinakumar H, Robinson M, Staud R, Berry RB, McCrae CS. Opioid use, pain intensity, age, and sleep architecture in patients with fibromyalgia and insomnia. Pain. 2019 Sep;160(9):2086-2092. doi: 10.1097/j.pain.0000000000001600. PMID 31180977
- [Derived] McCrae CS, Williams J, Roditi D, Anderson R, Mundt JM, Miller MB, Curtis AF, Waxenberg LB, Staud R, Berry RB, Robinson ME. Cognitive behavioral treatments for insomnia and pain in adults with comorbid chronic insomnia and fibromyalgia: clinical outcomes from the SPIN randomized controlled trial. Sleep. 2019 Mar 1;42(3):zsy234. doi: 10.1093/sleep/zsy234. PMID 30496533
- [Derived] Miller MB, Chan WS, Curtis AF, Boissoneault J, Robinson M, Staud R, Berry RB, McCrae CS. Pain intensity as a moderator of the association between opioid use and insomnia symptoms among adults with chronic pain. Sleep Med. 2018 Dec;52:98-102. doi: 10.1016/j.sleep.2018.08.015. Epub 2018 Sep 5. PMID 30296735
- [Derived] McCrae CS, Mundt JM, Curtis AF, Craggs JG, O'Shea AM, Staud R, Berry RB, Perlstein WM, Robinson ME. Gray Matter Changes Following Cognitive Behavioral Therapy for Patients With Comorbid Fibromyalgia and Insomnia: A Pilot Study. J Clin Sleep Med. 2018 Sep 15;14(9):1595-1603. doi: 10.5664/jcsm.7344. PMID 30176973
- [Derived] Curtis AF, Miller MB, Boissoneault J, Robinson M, Staud R, Berry RB, McCrae CS. Discrepancies in sleep diary and actigraphy assessments in adults with fibromyalgia: Associations with opioid dose and age. J Sleep Res. 2019 Oct;28(5):e12746. doi: 10.1111/jsr.12746. Epub 2018 Jul 31. PMID 30062746
- [Derived] Miller MB, Chan WS, Boissoneault J, Robinson M, Staud R, Berry RB, McCrae CS. Dynamic daily associations between insomnia symptoms and alcohol use in adults with chronic pain. J Sleep Res. 2018 Jun;27(3):e12604. doi: 10.1111/jsr.12604. Epub 2017 Sep 22. PMID 28940629